CLINICAL TRIAL: NCT00110760
Title: Randomized, Double-Blind, Placebo Controlled, Paired Study Evaluating S-Caine™ Peel (Lidocaine 7% and Tetracaine 7% Cream)for Induction of Local Dermal Anesthesia for Dermal Filler Injection on the Face of Adults
Brief Title: S-Caine™ Peel (Skin Numbing Cream) to Treat Pain During Skin Filler Injection in the Face
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCP-40-05
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-Caine Peel (Experimental)
  Interventions: Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%)
- Placebo Peel (Placebo Comparator)
  Interventions: Drug: Placebo Peel

INTERVENTIONS:
Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%) — S-Caine Peel was composed of a 1:1 eutectic mixture of 7% lidocaine and 7% tetracaine and was applied topically. S-Caine Peel was applied with a uniform thickness of approximately 1 mm and remained on the treatment area for 30 minutes (+/- 2 minutes).
  Other Names: Pliaglis
  Arms: S-Caine Peel
Drug: Placebo Peel — Placebo Peel applied topically with a uniform thickness of approximately 1 mm and remained on the treatment area for 30 minutes (+/- 2 minutes).
  Other Names: Placebo
  Arms: Placebo Peel

SUMMARY:
Injection of dermal filler is used as an aesthetic treatment to fill in unwanted wrinkles and scars. There can be substantial pain associated with dermal filler injections. For this reason, local anesthesia is often used to eliminate or minimize the pain. This anesthesia can be administered by injection or through the use of topical creams and ointments.

S-Caine™ Peel (lidocaine 7% and tetracaine 7% cream) is a eutectic formulation of lidocaine and tetracaine. The purpose of this study is to evaluate if S-Caine Peel is effective in providing topical local dermal anesthesia for dermal filler injections in adults.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo controlled, paired study to evaluate the efficacy of S-Caine Peel for local dermal anesthesia for facial dermal filler injection in 70 adults. The study was multi-center, with 3 centers participating.

Patients who presented to the study center for a dermal filler injection procedure and who met study entry criteria were invited to participate in the study. At the screening visit, the study, including potential risks and benefits, was clearly explained to each patient. A written and dated informed consent was obtained from each patient. A medical history was obtained including skin type, demographic data, and the use of concomitant medications. A brief physical examination was performed (a skin examination at the study treatment area and basic vital signs), and a urine pregnancy test was obtained for females of childbearing potential.

At the procedure visit, patients who met the eligibility criteria were assigned the lowest available sequential patient number. The randomization determined the placement of the S-Caine Peel and placebo with the active study drug applied to either the "top/right" or "bottom/left" treatment area and the placebo applied to the alternate treatment area. The treatment areas were defined as 2 similar anatomical locations that required similar amounts of dermal filler (as measured in mLs injected, and number of injections) administered. The point of reference for these designations was the patient's right and left or top and bottom. Patients had a concurrent administration of the study drugs, with the appropriate study drug applied to the top/right treatment area first followed immediately by the other study drug applied to the bottom/left treatment area. Study drug application was double-blind. The study drugs were applied with a uniform thickness of approximately 1 mm and remained on the skin for 30 minutes (+/- 2 minutes).

Upon removal of the study drugs (top/right treatment area removed first, followed immediately by removal of the other study drug from bottom/left treatment area), the investigator evaluated the treatment areas for erythema, edema, blanching and any adverse skin reaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient elects to undergo dermal filler injection in the face

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient has participated in a clinical trial of an unapproved drug within the previous 30 days
* Patient has participated in any previous clinical trial involving S-Caine Peel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 30 minutes
  Patient's evaluation of procedural pain intensity using the VAS. Immediately after completion of the dermal filler injections in each treatment area, patients completed a 100 mm horizontal VAS where 0 mm = no pain and 100 mm = the worst pain you can imagine

SECONDARY OUTCOMES:
Number of participants with adverse events | 30 minutes
  To monitor the nature and frequency of adverse events (AEs) associated with the use of S-Caine Peel
Patient's evaluation of the adequacy of pain relief | 30 minutes
  After the dermal filler procedure, each patient was asked to evaluate the efficacy of each study drug by answering the following questions: (i) Did this study drug provide adequate pain relief for the procedure (yes/no)? ; (ii) Would you have topical anesthesia administered using this study drug again if given the option (yes/no)?

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, MD, Principal Investigator — Tennessee Clinical Research Center
Locations (3):
- United States (3):
  - AboutSkin Dermatology, Englewood, Colorado
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - J&S Studies, Inc., Bryan, Texas